CLINICAL TRIAL: NCT03238079
Title: A Prospective, Open-Label, Multicenter Study of the Efficacy, Safety, Tolerability, and Pharmacokinetics of Therapure PlasmaCap IG in Adults and Children With Primary Immune Deficiency Diseases
Brief Title: Study of PlasmaCap IG in Adults and Children With PIDD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Therapure Biopharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBI-001-IGIV
Record Dates: First submitted 2017-07-21; First posted 2017-08-03 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Primary Immune Deficiency Diseases (PIDD)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label 10% IGIV (Experimental): IMP will be administered every 21 or 28 days in accordance with the subject's weekly regimen at screening for a period of 12 months. Subjects on a 21-day regimen will receive approximately 17 infusions, and subjects on a 28-day regimen will receive approximately 13 infusions.
  The starting dose will be the previous IGIV dose or a dose calculated from the previous SCIG dose up to a maximum of 900 mg/kg/mo.
  Interventions: Biological: 10% IGIV

INTERVENTIONS:
Biological: 10% IGIV — 300-900 mg/kg
  Other Names: Human Immunoglobulin

SUMMARY:
The purpose of this study is to investigate the efficacy, safety, tolerability, and pharmacokinetic profile of the investigational medicinal product (IMP) and to determine, on the basis of historical control data, how it compares with other 10% intravenous immunoglobulin (IGIV) products currently licensed in North America for the treatment of subjects with primary immune deficiency diseases (PIDD).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed clinical diagnosis of a PIDD, which requires treatment with IGIV:
* Subject/guardian has provided written informed consent (and assent, as applicable).
* Subject is between the ages of 2 and 70 years.
* Subject has received regular IGIV therapy at 21- or 28-day (±4 days) intervals for at least three consecutive months at a dose between 300-900 mg/kg/month prior to Screening or;
* Subject has received commercial SCIG at a dose of 300-900 mg/kg/month on any dosing schedule for at least 12 consecutive weeks prior to Screening. Subjects on SCIG must have received and tolerated IGIV treatment prior to SCIG treatment.
* Subject has a documented trough of ≥500 mg/dL in the 6 months prior to screening.
* Females of childbearing potential must be willing to use an effective form of birth control (eg, oral contraceptives) for the duration of the study, per IRB/REB guidelines.
* Subject agrees to comply with the requirements of the protocol.

Exclusion Criteria:

* Subject has secondary immunodeficiency.
* Subject has history of thrombotic events, such as deep vein thrombosis, myocardial infarction, cerebrovascular accident, pulmonary embolism, etc within the year prior to screening.
* Subject has had an immune globulin associated arterial or venous thrombotic/thromboembolic event (TEE) within 7 days of infusion or a TEE that is not associated with an immune globulin within one year of screening.
* Subject has received blood products (except for IGIV, SCIG, or albumin) within 6 months of screening.
* Subject has anemia (≤8.5 g/dL).
* Subject has levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3.0 times the upper limit of normal (ULN).
* Subject has severe neutropenia (≤1000 neutrophils per mm3).
* Subject is receiving other immunosuppressive or immunomodulatory drugs or chemotherapy.
* Subject is taking or has taken within the four weeks prior to screening prednisone at ≥0.15 mg/kg/day for more than 10 days.
* Subject has ever had a severe anaphylactic reaction to a blood or IgG product.
* Subject has lymphoid malignancy, leukemia, or any other history of malignancy within the past five years, except squamous cell or basal cell carcinoma of the skin (not melanoma).
* Subject has hypoalbuminemia, protein-losing enteropathy, or proteinuria greater than 300 mg/24 hours except for subjects with documented orthostatic proteinuria.
* Subject has immunoglobulin A (IgA) deficiency with known antibodies to IgA.
* Female who is pregnant, breastfeeding, or planning a pregnancy during the course of the study (women who become pregnant during the study will be withdrawn from the study).
* Any condition that is likely to interfere with evaluation of IMP or satisfactory conduct of the trial in the PI's opinion.
* Subjects who may not be compliant or have a history of non-compliance in the opinion of the PI.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-08-25 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean acute Serious Bacterial Infection (SBI) rate | 1 year
  The primary efficacy objective of the study is to demonstrate the efficacy of the IMP by determining that the mean annual acute SBI rate (as defined in Appendix 20.1) is statistically significantly lower than one infection per subject per year.

SECONDARY OUTCOMES:
Immunoglobulin G (IgG) trough concentration | up to 12 months per subject
  The average serum total IgG trough concentrations prior to each infusion
Days unable to perform daily activities | up to 12 months per subject
  The number of days unable to perform daily activities
Therapeutic IgG levels | up to 12 months per subject
  The ability of the IMP to maintain stable, therapeutic IgG levels

CONTACTS AND LOCATIONS:
Overall Officials: Mark Krause, Study Director — Therapure Biopharma
Locations (12):
- United States (11):
  - University of California, Los Angeles, California
  - IMMUNOe Health & Research Centers, Centennial, Colorado
  - University of South Florida, Tampa, Florida
  - Allergy Associates of the Palm Beaches, P.A., West Palm Beach, Florida
  - Institute for Asthma and Allergy, PC, Chevy Chase, Maryland
  - Optimed Research Ltd., Little Silver, New Jersey
  - Optimed Research LTD, Columbus, Ohio
  - Allergy Partners of North Texas, Dallas, Texas
  - AARA Research Center, Dallas, Texas
  - AAICPA, Irving, Texas
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- CHU Ste-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No